CLINICAL TRIAL: NCT01111981
Title: Safety and Efficacy of Clobetasol Propionate 0.05% E Foam in the Treatment of Central Centrifugal Cicatricial Alopecia
Brief Title: Safety and Efficacy of Clobetasol Propionate 0.05% E Foam in Alopecia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Callender Center for Clinical Research (Other)
Responsible Party: Valerie Callender, M.D., Callender Center for Clinical Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VDC2009O
Record Dates: First submitted 2010-04-26; First posted 2010-04-28 (Estimated); Last update posted 2010-04-28 (Estimated); Status verified 2010-04

CONDITIONS: Alopecia
Keywords: alopecia; CCCA - Central Centrifugal Cicatricial Alopecia
MeSH Terms: conditions — Alopecia | interventions — Clobetasol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Clobetasol Propionate 0.05% Emollient Foam — Clobetasol Propionate 0.05% E Foam to be applied to affected area once a day for 16 weeks
  Other Names: Olux-E

SUMMARY:
The purpose of this study is to ascertain the safety and efficacy of

Clobetasol Propionate 0.05% E Foam in the treatment of Central Centrifugal

Cicatricial Alopecia.

DETAILED DESCRIPTION:
Central Centrifugal Cicatricial Alopecia (CCCA) is an inflammation-induced

hair loss starting in the central scalp and progressing centrifugally. The

cause of CCCA is unknown. Early diagnosis and treatment is essential to stop

or slow the progression of scarring and permanent hair loss. Once scarring

occurs, the hair follicles are obliterated and the hair cannot regrow. Thus,

anti-inflammatory medications are used to decrease inflammation. Current

treatment includes topical and intralesional corticosteroids, oral

antibiotics, and hair transplantation, all which may take months to years to

show improvement. There is no evidence-based medicine on how to treat

primary cicatricial alopecias. Clobestasol Propionate 0.05% Emollient Foam is

an FDA-approved and marketed topical corticosteroid for the treatment of the

inflammatory and pruritic manifestations of moderate to severe corticosteroid-

responsive dermatoses of the scalp. Many studies found the foam to be less

irritating than the original formulation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CCCA, treated or untreated
* Score 0 - 1 on Scale/Questionnaire
* 18 years of age or older
* Women of African descent

Exclusion Criteria:

* Score > 1 on Scale/Questionnaire
* Alopecias other than CCCA, including alopecia arreata, lichen planopilaris, trichotillomania, and traction alopecia
* History of hair transplantation
* Children less than 18 years of age
* Males
* Women of non-African descent
* Pregnancy or breastfeeding. Women of childbearing age must use reliable forms of contraception (e.g., abstinence, oral contraceptives, or spermicide and condoms)
* Anti-dandruff shampoo within 30 days
* Anti-inflammatory medications such as antibiotics (doxycycline, minocycline, rifampin, etc.), steroids (oral prednisone, topical corticosteroids,etc.), NSAIDs (ibuprofen, aspirin, etc.)

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-02 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
Improvement of pruritis, tenderness, and pain | 4 months

SECONDARY OUTCOMES:
Absence of inflammation on biopsy | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Callender, M.D., Principal Investigator — Callender Skin for Clinical Research; Cherie Young, M.D., Study Director — Callender Center for Clinical Research
Locations (1):
- Callender Center for Clinical Research, Mitchellville, Maryland, United States

REFERENCES:
- [Derived] Callender VD, Kazemi A, Young CM, Chappell JA, Sperling LC. Safety and Efficacy of Clobetasol Propionate 0.05% Emollient Foam for the Treatment of Central Centrifugal Cicatricial Alopecia. J Drugs Dermatol. 2020 Jul 1;19(7):719-724. doi: 10.36849/JDD.2020.5201. PMID 32726554